CLINICAL TRIAL: NCT07046325
Title: Comparison Between Dexametidomedine\Bupivacaine and Plain Bupivacaine in Superior Trunk Block for Arthroscopic Shoulder Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FMASU R112/2025
Record Dates: First submitted 2025-06-15; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: Post Operative Pain, Acute; Arthroscopic Shoulder Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group B (Active Comparator): group administered Ultrasound guided STB with bupivacaine
  Interventions: Drug: Bupivacain
- group DB (Active Comparator): group administered Ultrasound guided STB with bupivacaine and dexametidomedine.
  Interventions: Drug: dexametedomidine; Drug: Bupivacain

INTERVENTIONS:
Drug: dexametedomidine — 1. Group DB: are administered Ultrasound guided STB with bupivacaine and dexametidomedine.
  Arms: group DB
Drug: Bupivacain — 2. Group B: are administered Ultrasound guided STB with bupivacaine.

SUMMARY:
Comparison between dexametidomedine\bupivacaine and plain bupivacaine in superior trunk block for arthroscopic shoulder surgeries

DETAILED DESCRIPTION:
This study will be conducted to investigate the efficacy of adding dexmedetomidine in STB for postoperative analgesia in patients undergoing arthroscopic shoulder surgery.

* Inclusion Criteria:

  1. age ;20-50 years old of both genders
  2. American Society of Anesthesiologists physical status I and II
  3. BMI less than 30
  4. Arthroscopic shoulder surgeries.
* Exclusion Criteria:

  1. Patients with ASA more than II
  2. Patients with a sepsis, malignancy anywhere
  3. Patient with bleeding tendencies or on anticoagulation therapy
  4. Patients with pre-existing neurologic deficit or neuropathy affecting brachial plexus
  5. Allergy to study drugs.

Study groups:

The patients will be randomized into 2 groups:

1. Group DB: are administered Ultrasound guided STB with bupivacaine and dexametidomedine.
2. Group B: are administered Ultrasound guided STB with bupivacaine.

Primary outcome:

Duration of analgesia of Superior trunck block.

Secondary outcome:

1. Cumulative dose of postoperative consumption of the rescue analgesia during 24h after STB
2. Durations of motor blockade (DOM)
3. Residual block related neurological symptoms
4. Hemodynamic variables
5. Dyspnea and sedation scale.

ELIGIBILITY:
Inclusion Criteria:

* Age ;20-50 years old
* Both genders
* American Society of Anesthesiologists physical status I and II
* BMI less than 30
* Arthroscopic shoulder surgeries.

Exclusion Criteria:

* Patients with ASA more than II
* Patients with a sepsis, malignancy anywhere
* Patient with bleeding tendencies or on anticoagulation therapy
* Patients with pre-existing neurologic deficit or neuropathy affecting brachial plexus
* Allergy to study drugs.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia of Superior trunck block. | 24 hours
  The DOA will be defined as the time interval between STB and the first need for the rescue analgesics.

CONTACTS AND LOCATIONS:
Overall Officials: fagr fathy abdo, Medical Doctorate, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt